CLINICAL TRIAL: NCT06933368
Title: A 12-Week, Randomized, Controlled, Examiner-blind, Clinical Study to Evaluate the Efficacy of a Cetylpyridinium Chloride Mouthwash in Improving Gingival Health and Reducing Plaque Accumulation
Brief Title: A Clinical Study to Evaluate the Efficacy of a Cetylpyridinium Chloride Mouthwash in Improving Gingival Health and Reducing Plaque Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300268
Record Dates: First submitted 2025-04-16; First posted 2025-04-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Products (Toothpaste + Mouthwash) (Experimental): Participants will be instructed to brush their teeth with the toothpaste (Crest Cavity Protection) for at least one minute twice daily (morning and evening) for 12 weeks. After each brushing, participants will swish 20 milliliter (ml) of experimental mouthwash for 30 seconds without rinsing with water after use of mouthwash.
  Interventions: Drug: Crest Cavity Protection Toothpaste; Drug: Experimental Mouthwash
- Reference Product (Toothpaste) (Active Comparator): Participants will be instructed to brush their teeth with the toothpaste (Crest Cavity Protection) for at least one minute twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Crest Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Crest Cavity Protection Toothpaste — Toothpaste containing 0.243% w/w NaF.
Drug: Experimental Mouthwash — Mouthwash containing 0.085% w/w CPC.
  Arms: Test Products (Toothpaste + Mouthwash)

SUMMARY:
The aim of this 12-week clinical study is to evaluate the ability of an experimental mouthwash, containing 0.085 percent (%) Cetylpyridinium chloride (CPC) as an adjunct to toothbrushing with a regular fluoride toothpaste, to improve gingival health and plaque accumulation compared to a regular fluoride toothpaste alone in participants with plaque-induced mild to moderate gingivitis.

DETAILED DESCRIPTION:
This will be a single-center, 12-week, randomized, controlled, single blind (examiner only), 2-treatment arms, parallel group, stratified (by sex [male/female]) study, investigating gingival health and subgingival plaque reduction on healthy participants after twice daily using of an experimental mouthwash containing 0.085% weight/weight (w/w) CPC in combination with a commercially available regular toothpaste containing 0.243% w/w Sodium Fluoride (NaF) compared to a commercially available regular toothpaste containing 0.243% w/w NaF with no known anti-gingivitis nor anti plaque efficacy properties as control group. Approximately 132 participants (approximately 66 per group) will be randomized to ensure approximately 120 evaluable participants (approximately 60 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is at least 18 years old, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant oral health that meets all the following:
* At screening (visit 1):

  1. Participant with at least 20 natural, permanent teeth.
  2. Participant with at least 40 evaluable surfaces for MGI, bleeding index (BI), and TPI.
  3. A participant with plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by a gross visual examination at the screening visit.
* At baseline (visit 2; prior to dental prophylaxis)

  1. A participant with 10% to 30% bleeding sites.
  2. A participant with overall TPI score >=1.5.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical, psychiatric condition or laboratory abnormality or any other clinical serious or unstable conditions (for example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who is a pregnant female (self-reported) or intending to become pregnant over the duration of the study.
* A female participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who is a current smoker or an ex-smoker (including vaping) who stopped within 6 months of Screening.
* A participant who is using smokeless forms of tobacco (for example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed with xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding (for example, type 2 diabetes).
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (for example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* Medication exclusions: At screening (Visit 1):

  1. A participant using any antibiotic medication within 4 weeks prior to screening or at any time during the study.
  2. A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
  3. A participant currently taking a systemic medication (for example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy or as a premedication requirement before an invasive examinations and prophylaxis (for example, knee replacement, Mitral valve prolapse etc.), which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  4. A participant who has used an antibacterial dentifrice or mouthwash (for example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, within 4 weeks prior to screening.
* Medication exclusions: At baseline (Visit 2):

  1. A participant who has taken (in the previous 4 weeks), any antibiotics.
  2. A participant who requires the need for antibiotic premedication prior to a dental prophylaxis or taking some blood thinning medication that prohibit the safe conduct of a dental cleaning. Note: Medical consultation may need to be obtained from participant's physician at the examiner's discretion.
  3. A participant who has taken (in the previous 4 weeks) a systemic medication (for example, anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy as a premedication requirement before an invasive examinations and prophylaxis (for example, knee replacement, Mitral valve prolapse etc.), which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  4. A participant who has used an antibacterial dentifrice or mouthwash (for example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, in the period between Screening and the Baseline visit.
* Periodontal exclusions:

  1. A participant who has more than three tooth sites with probing pocket depth >=4 mm.
  2. A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  3. A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
* Dental exclusions:

  1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  2. A participant who has dentures (partial or full).
  3. A participant who has an orthodontic appliance (bands, appliances, or fixed/ removable retainers).
  4. A participant who received orthodontic therapy within 3 months of Screening.
  5. A participant who has numerous restorations in a poor state of repair.
  6. A participant who has any dental condition (for example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  7. A participant who has had dental prophylaxis within 12 weeks of Screening.
  8. A participant who has had teeth bleaching within 12 weeks of Screening.
  9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Number of Bleeding Sites (Overall) At Week 12 | Week 12
  Gingival bleeding will be assessed according to the expanded bleeding index (EBI), by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) before recording the number of gingival units which bleed. The number of bleeding sites is calculated as the number of evaluable tooth sites (having 2/3rds of the natural tooth surface gradable for assessment) with bleeding observed immediately on probing or within 30 seconds of probing.

SECONDARY OUTCOMES:
Number of Bleeding Sites (Interproximal) At Week 12 | Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) before recording the number of gingival units which bleed. The number of bleeding sites is calculated as the number of evaluable tooth sites (having 2/3rds of the natural tooth surface gradable for assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Number of Bleeding Sites (Overall) At Week 6 | Week 6
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) before recording the number of gingival units which bleed. The number of bleeding sites is calculated as the number of evaluable tooth sites (having 2/3rds of the natural tooth surface gradable for assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Number of Bleeding Sites (Interproximal) At Week 6 | Week 6
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) before recording the number of gingival units which bleed. The number of bleeding sites is calculated as the number of evaluable tooth sites (having 2/3rds of the natural tooth surface gradable for assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Mean EBI (Overall) At Week 6 and Week 12 | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) and gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0= no bleeding after 30 seconds, 1= bleeding observed within 30 seconds of probing, 2=bleeding observed immediately on probing. Lower score indicates improvement in the symptoms.
Mean EBI (Interproximal) At Week 6 and Week 12 | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degree, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. All scorable teeth in one quadrant will be probed first (approximately 30 seconds) and gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0= no bleeding after 30 seconds, 1= bleeding observed within 30 seconds of probing, 2=bleeding observed immediately on probing. Lower score indicates improvement in the symptoms.
Mean Modified Gingival Index (MGI) (Overall) At Week 6 and Week 12 | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). The MGI will be assessed for all scorable teeth (second permanent molar to second permanent molar in each arch) by an appropriately qualified examiner using 5-point scoring system ranging from 0 to 4, where 0= Absence of inflammation, 1= Mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit, 2= Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit, 3= Moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit, 4= Severe inflammation; marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms of gingivitis.
Mean MGI (Interproximal) At Week 6 and Week 12 | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). The MGI will be assessed for all scorable teeth (second permanent molar to second permanent molar in each arch) by an appropriately qualified examiner using 5-point scoring system, where 0= Absence of inflammation, 1= Mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit, 2= Mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit, 3= Moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit, 4= Severe inflammation; marked redness, edema and/ or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms of gingivitis.
Mean Turesky Plaque Index (TPI) (Overall) at Week 6 and Week 12 | Week 6 and Week 12
  TPI will be used to assess plaque on all gradable teeth. The plaque will be disclosed using a plaque disclosing dye solution. The TPI will be assessed on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores should be recorded buccally/labially (distal, body, mesial sites) and three scores lingually/palatally (distal, body, mesial sites). Disclosed plaque will be scored using 6-point scale ranging from 0 to 5, where 0= No plaque, 1= Separate flecks of plaque at the cervical margin, 2= Thin continuous band of plaque (up to 1 millimeter [mm]) at the cervical margin, 3= Band of plaque wider than 1 mm but covering less than (<) 1/3 of the tooth surface, 4= Plaque covering more than or equal to (>=) 1/3 but < 2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement.
Mean TPI (Interproximal) at Week 6 and Week 12 | Week 6 and Week 12
  TPI will be used to assess plaque on all gradable teeth. The plaque will be disclosed using a plaque disclosing dye solution. The TPI will be assessed on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores should be recorded buccally/labially (distal, body, mesial sites) and three scores lingually / palatally (distal, body, mesial sites). Disclosed plaque will be scored using 6-point scale ranging from 0 to 5, where 0= No plaque, 1= Separate flecks of plaque at the cervical margin, 2= Thin continuous band of plaque (up to 1 mm) at the cervical margin, 3= Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4= Plaque covering >=1/3 but <2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trialregister@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.